CLINICAL TRIAL: NCT03352089
Title: Positron Emission Tomography / Magnetic Resonance Imaging in Aortic Stenosis
Acronym: PASS
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 17/SS/0066
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Aortic Stenosis; Transthyretin Amyloidosis
Keywords: Magnetic resonance imaging; Positron emission tomography
MeSH Terms: conditions — Aortic Valve Stenosis; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — lood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic stenosis group: Patients with severe aortic stenosis >70 years of age referred for aortic valve intervention
- Healthy volunteer group: Patients with no history of symptoms to suggest current cardiovascular disease >70 years of age

SUMMARY:
Aortic stenosis is the most common valve disease requiring surgery in the Western world. It is defined by progressive calcification and fibrosis of the valve leaflets and restricted valve opening. This in turn exposes the heart muscle (left ventricle) to increasing pressure leading to heart muscle thickening (left ventricular hypertrophy, LVH) to normalise wall stress and maintain heart output (stroke volume). The only treatment available is relief of pressure overload by surgical or minimally invasive valve replacement (TAVI).

Transthyretin (TTR) amyloidosis is a condition characterised by deposition of insoluble transthyretin protein (a small protein tetramer produced in the liver) in various tissues, predominantly in the heart. Although there are inherited forms caused by specific TTR gene mutations, most cases occur in older individuals with non-mutated TTR (wild-type). The finding of TTR plaques in elderly individuals is relatively common; in a post-mortem study 22-25% of patients over the age of 80 had evidence of cardiac amyloid deposition. However, there is significant progressive amyloid accumulation in a small percentage of individuals leading to heart muscle thickening and heart failure. No medical treatments are currently licensed although several agents are at advanced stages of clinical trials.

As both the above conditions are increasingly common in the elderly population and characterised by increased heart muscle thickening, there is the potential for them to coexist unrecognised in individual patients. The prevalence of cardiac amyloidosis in clinical populations with significant aortic stenosis is not known however small series have estimated somewhere in the region of 6-29%. Other data have suggested that patients with aortic stenosis and concurrent cardiac amyloidosis have an adverse prognosis even despite AVR. It is therefore important to identify aortic stenosis patients with coexistent amyloidosis both in terms of predicting prognosis and because it may influence decisions about whether to proceed to valve intervention.

PET/MR is an emerging technique, which combines the excellent temporal and spatial resolution of MRI with the sensitive molecular imaging of PET. PET/MR has significant advantages over PET/CT (the currently more widely used approach) in that it offers superior tissue characterisation, improved correction for cardiac and respiratory motion and major reductions in radiation exposure. Whilst there are concerns about its ability to provide reliable attenuation correction of the PET data, these issues appear to have been largely overcome with recent techniques proposed by our group. MR is also more naturally suited to the imaging of certain tissues in the body compared to CT including the left ventricular myocardium.

In aortic stenosis, MRI has become the gold-standard technique for examining the heart muscle (myocardium) with the unique ability to assess its tissue composition. In particular both late gadolinium enhancement (LGE) and T1 mapping based techniques are able to detect heart scarring (fibrosis) which act as biomarkers of left ventricular decompensation and are strongly associated with poor patient outcomes. CMR is also the gold-standard non-invasive technique for detecting cardiac amyloid, which is associated with both a characteristic pattern of LGE and high native T1 values. However it is not currently able to differentiate between the two different types of cardiac amyloid TTR and AL amyloidosis, which have different prognoses and treatments. Preliminary studies conducted by our group have suggested that 18F-NaF PET when added to CMR can make this distinction on the basis that this tracer binds to TTR deposits but not AL deposits, may be able to differentiate between the two. Importantly we have also used the same PET tracer as a marker of calcification activity in the aortic valve, demonstrating its ability to predict disease progression and cardiac events.

In this study, we will investigate whether PET/MR could be used as "one-stop" imaging in aortic stenosis in whom valve intervention is being considered to assess in detail functional and structural properties of both the valve and myocardium and identify cases of significant cardiac TTR amyloid deposition.

ELIGIBILITY:
Inclusion Criteria (AS group)

* Severe aortic stenosis
* Referred for aortic valve intervention (surgical AVR / TAVI)
* High clinical suspicion of amyloid (e.g. low-flow low-gradient AS, inappropriate LVH)
* Age >70 years
* Willing and able to comply with study protocol

Exclusion Criteria (AS group)

* Inability to give informed consent
* Contraindication to MRI scanning (e.g. permanent pacemaker)
* Significant renal impairment (eGFR <30 ml/min/1.73 m2)
* Coexistent moderate or severe aortic regurgitation or mitral stenosis
* Acute valvular heart disease (e.g. acute mitral regurgitation or endocarditis)
* Acute pulmonary oedema or cardiogenic shock

Inclusion Criteria (Healthy volunteers)

* No symptoms suggesting current cardiovascular disease
* Age >70
* Willing and able to comply with study protocol

Exclusion Criteria (Healthy volunteers)

* Inability to give informed consent
* Contraindication to MRI scanning (e.g. permanent pacemaker)
* Significant renal impairment (eGFR <30 ml/min/1.73 m2)
* Known significant valvular heart disease (more than mild regurgitant valve lesion or any stenotic lesion)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: AS group: patients at NHS Lothian referred for aortic valve intervention
  Healthy volunteer group: healthy volunteers from South-East Scotland who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
PET signal intensity quantified by calculation of standard uptake values | Pre surgery scan

CONTACTS AND LOCATIONS:
Overall Officials: Russell J Everett, MBBS, Principal Investigator — University of Edinburgh / NHS Lothian
Locations (1):
- University of Edinburgh / NHS Lothian, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided